CLINICAL TRIAL: NCT01171625
Title: Carpentier-Edwards PERIMOUNT Magna Ease Pericardial Bioprosthesis in the Aortic Position, Model 3300TFX
Brief Title: Carpentier-Edwards PERIMOUNT Magna Ease Pericardial Bioprosthesis, Model 3300TFX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-08
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease; Aortic Valve Disorder; Heart Failure; Aortic Valve Stenosis; Aortic Valve Insufficiency
Keywords: PERIMOUNT, Aortic valve replacement/regurgitation
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease; Heart Failure; Aortic Valve Stenosis; Aortic Valve Insufficiency; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CEP Aortic Bioprothesis, model 3300TFX (Other)
  Interventions: Device: Implantation of CEP Magna Ease Model 3300TFX

INTERVENTIONS:
Device: Implantation of CEP Magna Ease Model 3300TFX — Heart Valve Surgery
  Other Names: CEP Magna Ease MOdel 3300TFX

SUMMARY:
The purpose of the study is to demonstrate the long term safety and effectiveness of the Carpentier-Edwards PERIMOUNT Magna Ease Valves in patients undergoing aortic valve replacement with or without concomitant procedures requiring cardiopulmonary bypass.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, interventional study to be conducted in the US and outside the US (OUS). This study will enroll a minimum of 225 patients implanted with the study valve in order to achieve 101 aortic valve replacement subjects each followed for a minimum of 8 years. The study will include male and female patients, 18 years or older, requiring replacement for a diseased, damaged or malfunctioning natural or prosthetic aortic valve. Patients will be followed and assessed after implant at discharge, 6 months, one year, and annually for a minimum of 8 years.

ELIGIBILITY:
Inclusion Criteria:

1. The patient requires, as indicated in the preoperative evaluation, a replacement aortic valve.
2. The patient is an average or better operative risk.
3. The patient is geographically stable and agrees to attend follow-up assessments at the hospital of surgical services for at least 8 years.
4. The patient is 18 years or older.
5. The patient has signed and dated the subject informed consent form prior to surgery.

Exclusion Criteria:

1. The patient has any known non-cardiac life-threatening disease, which will limit the patient's life expectancy below 1 year.
2. The patient presents with active endocarditis within the last 3 months.
3. The patient has an abnormal calcium metabolism (e.g., chronic renal failure, hyperparathyroidism).
4. The patient has an aneurismal aortic degenerative condition (e.g., cystic medial necrosis, Marfan's syndrome).
5. The patient is pregnant or lactating.
6. The patient is an intravenous drug abuser.
7. The patient is currently a prison inmate.
8. The patient is currently participating in a study of an investigational drug or device.
9. The patient requires replacement of a native or prosthetic mitral, tricuspid or pulmonic valve.
10. The patient requires a repair of the mitral or tricuspid valve with the use of an annuloplasty device.
11. The patient was previously enrolled in the study.
12. The patient had a prior mitral, tricuspid or pulmonic valve surgery, which included implantation of a bioprosthetic valve, mechanical valve, or annuloplasty ring that will remain in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - Mercy General Hospital, Sacramento, California
  - Cooper University Hospital, Camden, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Providence Heart & Vascular Institute, Portland, Oregon
  - St. Marks Hospital, Salt Lake City, Utah
- Universitatslinik fur Chirurgie, Innsbruck, Austria
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Paul's Hospital, Vancouver
- Germany (2):
  - Liknik fur Herz und BefaBchirurgie Im Deuschen Herzzentrum, Munich, Lazarettstr
  - Klinik fur Herz-, Thorax-, Transplantations- und Gefabchirurgie, Hanover
- Hospital Peutra de Hierro, San Martin de Porres 4, Madrid, Spain
- United Kingdom (2):
  - Papworth Hospital NHS foundation Trust, Papworth Everard, Cambridge
  - Blackpool Victoria Hospital, Blackpool, Lancashire

REFERENCES:
- [Result] Wahlers TCW, Andreas M, Rahmanian P, Candolfi P, Zemanova B, Giot C, Ferrari E, Laufer G. Outcomes of a Rapid Deployment Aortic Valve Versus Its Conventional Counterpart: A Propensity-Matched Analysis. Innovations (Phila). 2018 May/Jun;13(3):177-183. doi: 10.1097/IMI.0000000000000509. PMID 29912142
- See also: New York Heart Association Classification — https://www.heart.org/en/health-topics/heart-failure/what-is-heart-failure/classes-of-heart-failure

RESULTS

PARTICIPANT FLOW:
Groups:
- Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX: Subjects who received the Carpentier-Edwards® PERIMOUNT® Magna Ease™ valve, Model 3300TFX, undergoing isolated aortic valve replacement.
Period: Overall Study
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Started | 283
Subjects Implanted With Device | 258
Completed | 103
Not Completed | 180
Not completed — On-Protocol | 67
Not completed — Death | 38
Not completed — Withdrawal by Subject | 31
Not completed — Explanted | 10
Not completed — Lost to Follow-up | 5
Not completed — Patient received valve-in-valve | 3
Not completed — Other | 1
Not completed — Consented but did not receive device | 25

BASELINE CHARACTERISTICS:
Population: The outcome is reported for subjects who received the Carpentier-Edwards PERIMOUNT Magna Ease, Model 3300TFX, device where data is available.
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 167
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subject's Percentage of Long Term Safety Performance
Description: Long term safety performance will be evaluated by comparing the linearized yearly rates to the objective performance criteria (OPC) referenced in the Food and Drug Administration (FDA) 1994 Draft Heart Valve Guidance.
  Expressed as the Number of late events divided by the total number of late patient years times 100. Late patient years are calculated from 31 days post-implant to the date of the last contact (follow up or adverse event).
Time Frame: 31 days through 8 years post-implant
Population: as for baseline characteristics
Measure: Number; unit: Percentage of events/late patient years
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
Percentage of events/late patient years
  Thromboembolism | 1.5
  All Hemorrhage | 2.7
  All Perivalvular Leak | 0.2
  Endocarditis | 0.4

2. Primary Outcome: Number of Subject's in NYHA Functional Class I or II at 8 Year Post-Implant
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
Time Frame: 8 years post-implant
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 98
Participants
  Class I | 57
  Class II | 35

3. Primary Outcome: Subject's New York Heart Association (NYHA) Functional Class at 8 Years Post-Implant Compared to Baseline
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: 8 Years post-implant
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 97
Participants
  Improve | 60
  Same | 31
  Worse | 6

4. Secondary Outcome: Percent of Early Adverse Events
Description: Number of early adverse events occurring within 30 days of procedure divided by the number of enrolled subjects times 100.
Time Frame: Events occurring within 30 days of procedure
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Early Adverse Events
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
Percentage of Early Adverse Events
  Bleeding Event | 6.2
  Major Bleeding Event | 5.0
  Thromboembolism | 1.9
  Endocarditis | 0.0
  Structural Valve Deterioration | 0.0
  Reoperation Due to SVD | 0.0
  Hemolysis | 0.0
  Non-Structural Valve Deterioration | 0.4
  Perivalvular Leak | 0.4
  Major Perivalvular Leak | 0.4
  Valve Thrombosis | 0.0
  Explant | 1.2
  Death | 0.4
  Valve-related death | 0.0

5. Secondary Outcome: Percentage of Late Adverse Events
Description: Number of late events divided by the total number of late patient years times 100. Late patient years are calculated from 31 days post-implant to the date of the last contact (follow up or adverse event).
Time Frame: Events occurring >= 31 days and up through 8 years post-implant
Population: as for baseline characteristics
Measure: Number; unit: Percentage of events/late patient years
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
Percentage of events/late patient years
  Bleeding Event | 2.7
  Major Bleeding Event | 1.3
  Thromboembolism | 1.5
  Endocarditis | 0.4
  Structural Valve Deterioration | 1.0
  Reoperation Due to SVD | 0.6
  Hemolysis | 0.1
  Non-Structural Valve Deterioration | 0.3
  Perivalvular Leak | 0.2
  Major Perivalvular Leak | 0.1
  Valve Thrombosis | 0.0
  Explant | 0.5
  Death | 2.3
  Valve-related death | 0.5

6. Secondary Outcome: Percent of Subjects With Freedom From Serious Adverse Events (SAE) Post-implant > 30 Days
Description: Subject's freedom from Serious Adverse Events at > 30 days post-implant. Time to events were estimated by Kaplan-Meier method.
Time Frame: 1 Year, 2 Years, 3 Years, 4 Years, 5 Years, 6 Years, 7 Years, and 8 Years post-implant
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Magna Ease™, Model 3300TFX - 1 Year Post-Implant; Magna Ease™, Model 3300TFX - 2 Year Post-Implant; Magna Ease™, Model 3300TFX - 3 Year Post-Implant; Magna Ease™, Model 3300TFX - 4 Year Post-Implant; Magna Ease™, Model 3300TFX - 5 Year Post-Implant; Magna Ease™, Model 3300TFX - 6 Year Post-Implant; Magna Ease™, Model 3300TFX - 7 Year Post-Implant; Magna Ease™, Model 3300TFX - 8 Year Post-Implant: Subjects who received the Carpentier-Edwards® PERIMOUNT® Magna Ease™ valve, Model 3300TFX, undergoing isolated aortic valve replacement.
Arm/Group | Magna Ease™, Model 3300TFX - 1 Year Post-Implant | Magna Ease™, Model 3300TFX - 2 Year Post-Implant | Magna Ease™, Model 3300TFX - 3 Year Post-Implant | Magna Ease™, Model 3300TFX - 4 Year Post-Implant | Magna Ease™, Model 3300TFX - 5 Year Post-Implant | Magna Ease™, Model 3300TFX - 6 Year Post-Implant | Magna Ease™, Model 3300TFX - 7 Year Post-Implant | Magna Ease™, Model 3300TFX - 8 Year Post-Implant
Number analyzed (Participants) | 258 | 258 | 258 | 258 | 258 | 258 | 258 | 258
percentage of subjects
  Death | 97.60 [95.71 to 99.50] | 97.19 [95.14 to 99.24] | 95.50 [92.89 to 98.10] | 93.76 [90.70 to 96.82] | 91.54 [87.98 to 95.09] | 89.20 [85.18 to 93.21] | 85.16 [80.34 to 89.98] | 80.69 [74.94 to 86.43]
  Valve-related death | 99.60 [98.83 to 100.0] | 99.60 [98.83 to 100.0] | 98.74 [97.32 to 100.0] | 98.28 [96.61 to 99.95] | 97.81 [95.91 to 99.71] | 97.31 [95.18 to 99.44] | 96.66 [94.19 to 99.13] | 95.79 [92.81 to 98.77]
  Reoperation | 97.63 [95.76 to 99.51] | 97.21 [95.18 to 99.25] | 96.78 [94.59 to 98.98] | 95.89 [93.39 to 98.39] | 95.89 [93.39 to 98.39] | 95.37 [92.69 to 98.06] | 94.07 [90.87 to 97.27] | 89.83 [85.09 to 94.58]
  Explant | 98.04 [96.34 to 99.74] | 97.62 [95.74 to 99.50] | 97.19 [95.14 to 99.25] | 96.30 [93.92 to 98.68] | 96.30 [93.92 to 98.68] | 96.30 [93.92 to 98.68] | 95.65 [92.96 to 98.33] | 94.81 [91.70 to 97.93]
  Bleeding Event | 88.44 [84.48 to 92.40] | 86.76 [82.55 to 90.98] | 84.13 [79.55 to 88.71] | 83.22 [78.51 to 87.92] | 81.79 [76.90 to 86.69] | 81.29 [76.33 to 86.25] | 80.63 [75.54 to 85.72] | 77.95 [72.20 to 83.70]
  Major Bleeding Event | 92.51 [89.26 to 95.75] | 92.09 [88.75 to 95.42] | 90.33 [86.64 to 94.02] | 90.33 [86.64 to 94.02] | 88.91 [84.95 to 92.87] | 88.40 [84.34 to 92.47] | 87.75 [83.52 to 91.98] | 85.08 [80.02 to 90.15]
  Thromboembolism | 96.03 [93.61 to 98.44] | 94.32 [91.43 to 97.22] | 92.56 [89.25 to 95.88] | 92.11 [88.69 to 95.52] | 90.70 [86.98 to 94.41] | 89.68 [85.75 to 93.62] | 88.39 [84.13 to 92.66] | 86.68 [81.88 to 91.47]
  Endocarditis | 98.81 [97.47 to 100.0] | 98.39 [96.83 to 99.96] | 98.39 [96.83 to 99.96] | 97.94 [96.15 to 99.73] | 97.94 [96.15 to 99.73] | 97.94 [96.15 to 99.73] | 97.27 [95.07 to 99.48] | 97.27 [95.07 to 99.48]
  Perivalvular leak | 98.78 [97.41 to 100.0] | 98.36 [96.77 to 99.95] | 98.36 [96.77 to 99.95] | 98.36 [96.77 to 99.95] | 98.36 [96.77 to 99.95] | 98.36 [96.77 to 99.95] | 98.36 [96.77 to 99.95] | 98.36 [96.77 to 99.95]
  Major perivalvular leak | 99.20 [98.09 to 100.0] | 99.20 [98.09 to 100.0] | 99.20 [98.09 to 100.0] | 99.20 [98.09 to 100.0] | 99.20 [98.09 to 100.0] | 99.20 [98.09 to 100.0] | 99.20 [98.09 to 100.0] | 99.20 [98.09 to 100.0]
  Hemolysis | 99.18 [98.04 to 100.0] | 99.18 [98.04 to 100.0] | 99.18 [98.04 to 100.0] | 99.18 [98.04 to 100.0] | 99.18 [98.04 to 100.0] | 99.18 [98.04 to 100.0] | 99.18 [98.04 to 100.0] | 99.18 [98.04 to 100.0]
  Non-structural valve dysfunction | 98.78 [97.41 to 100.0] | 98.36 [96.77 to 99.95] | 98.36 [96.77 to 99.95] | 97.91 [96.09 to 99.73] | 97.91 [96.09 to 99.73] | 97.91 [96.09 to 99.73] | 97.91 [96.09 to 99.73] | 97.91 [96.09 to 99.73]
  Structural valve deterioration | 100.0 [100.0 to 100.0] | 99.57 [98.74 to 100.0] | 99.13 [97.94 to 100.0] | 99.13 [97.94 to 100.0] | 99.13 [97.94 to 100.0] | 97.07 [94.75 to 99.39] | 95.74 [92.81 to 98.67] | 90.08 [84.74 to 95.42]
  Valve thrombosis | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

7. Secondary Outcome: Subject's Average Peak Systolic Gradient (mmHg) Measurements at 8 Years Post-implant
Description: Peak systolic gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury. The data summary will be stratified by valve size.
Time Frame: 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 89
mmHg
  19 mm: number analyzed (Participants) | 4
  19 mm | 24.6 (17.94)
  21 mm: number analyzed (Participants) | 11
  21 mm | 24.7 (23.52)
  23 mm: number analyzed (Participants) | 33
  23 mm | 26.3 (21.41)
  25 mm: number analyzed (Participants) | 35
  25 mm | 21.6 (8.94)
  27 mm: number analyzed (Participants) | 4
  27 mm | 22.1 (8.81)
  29 mm: number analyzed (Participants) | 2
  29 mm | 23.1 (15.41)

8. Secondary Outcome: Subject's Average Mean Systolic Gradient (mmHg) Measurements at 8 Years Post-implant.
Description: Mean systolic gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Mean gradient values depend on the size and type of valve. The data summary will be stratified by valve size.
Time Frame: 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 89
mmHg
  19 mm: number analyzed (Participants) | 4
  19 mm | 17.7 (6.38)
  21 mm: number analyzed (Participants) | 11
  21 mm | 17.2 (10.82)
  23 mm: number analyzed (Participants) | 33
  23 mm | 16.2 (10.46)
  25 mm: number analyzed (Participants) | 35
  25 mm | 12.7 (4.56)
  27 mm: number analyzed (Participants) | 4
  27 mm | 12.2 (4.51)
  29 mm: number analyzed (Participants) | 2
  29 mm | 13.3 (9.48)

9. Secondary Outcome: Subject's Average Effective Orifice Area Measurements at 8 Years Post-implant.
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the aortic valve. The data summary will be stratified by valve size.
Time Frame: 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Centimeters Squared
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 86
Centimeters Squared
  19 mm: number analyzed (Participants) | 3
  19 mm | 1.0 (0.15)
  21 mm: number analyzed (Participants) | 11
  21 mm | 1.4 (0.40)
  23 mm: number analyzed (Participants) | 33
  23 mm | 1.4 (0.53)
  25 mm: number analyzed (Participants) | 34
  25 mm | 1.7 (0.47)
  27 mm: number analyzed (Participants) | 3
  27 mm | 2.1 (0.32)
  29 mm: number analyzed (Participants) | 2
  29 mm | 1.9 (0.44)

10. Secondary Outcome: Subject's Average Effective Orifice Area Index (EOAI) Measurements at 8 Years Post-implant.
Description: Effective orifice area index represents the minimal cross-sectional area of the blood flow downstream of the aortic valve divided by the person's body surface area. The data summary will be stratified by valve size.
Time Frame: 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: centimeters squared/meters squared
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 86
centimeters squared/meters squared
  19 mm: number analyzed (Participants) | 3
  19 mm | 0.6 (0.11)
  21 mm: number analyzed (Participants) | 11
  21 mm | 0.7 (0.20)
  23 mm: number analyzed (Participants) | 33
  23 mm | 0.8 (0.32)
  25 mm: number analyzed (Participants) | 34
  25 mm | 0.8 (0.21)
  27 mm: number analyzed (Participants) | 3
  27 mm | 1.1 (0.10)
  29 mm: number analyzed (Participants) | 2
  29 mm | 0.9 (0.24)

11. Secondary Outcome: Subject's Average Performance Index Measurements at 8 Years Post-implant.
Description: Performance index is defined as the subject's effective orifice area (the cross-sectional area of the blood flow downstream of the aortic valve) divided by the subject's native orifice area. The data summary will be stratified by valve size.
Time Frame: 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: cm^2/cm^2
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 86
cm^2/cm^2
  19 mm: number analyzed (Participants) | 3
  19 mm | 0.5 (0.09)
  21 mm: number analyzed (Participants) | 11
  21 mm | 0.5 (0.14)
  23 mm: number analyzed (Participants) | 33
  23 mm | 0.4 (0.18)
  25 mm: number analyzed (Participants) | 34
  25 mm | 0.4 (0.10)
  27 mm: number analyzed (Participants) | 3
  27 mm | 0.4 (0.04)
  29 mm: number analyzed (Participants) | 2
  29 mm | 0.3 (0.09)

12. Secondary Outcome: Subject's Average Cardiac Output Measurements at 8 Years Post-implant.
Description: The amount of blood the heart pumps through the circulatory system in a minute. The data summary will be stratified by valve size.
Time Frame: 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 86
Liters per minute
  19 mm: number analyzed (Participants) | 3
  19 mm | 3.6 (0.32)
  21 mm: number analyzed (Participants) | 11
  21 mm | 5.2 (1.23)
  23 mm: number analyzed (Participants) | 33
  23 mm | 5.0 (1.10)
  25 mm: number analyzed (Participants) | 34
  25 mm | 5.1 (1.28)
  27 mm: number analyzed (Participants) | 3
  27 mm | 6.3 (2.10)
  29 mm: number analyzed (Participants) | 2
  29 mm | 5.3 (0.78)

13. Secondary Outcome: Subject's Average Cardiac Index Measurements at 8 Years Post-implant.
Description: Cardiac index is an assessment that divides the cardiac output from left ventricle in one minute by the person's body surface area (BSA), thus relating heart performance to the size of the individual. The data summary will be stratified by valve size.
Time Frame: 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 86
L/min/m^2
  19 mm: number analyzed (Participants) | 3
  19 mm | 2.3 (0.22)
  21 mm: number analyzed (Participants) | 11
  21 mm | 2.9 (0.55)
  23 mm: number analyzed (Participants) | 33
  23 mm | 2.7 (0.60)
  25 mm: number analyzed (Participants) | 34
  25 mm | 2.6 (0.60)
  27 mm: number analyzed (Participants) | 3
  27 mm | 3.1 (0.91)
  29 mm: number analyzed (Participants) | 2
  29 mm | 2.6 (0.32)

14. Secondary Outcome: Subject's Amount of Aortic Valvular Regurgitation at 8 Years Post-Implant.
Description: Aortic valvular regurgitation occurs when the aortic valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Aortic valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation.
Time Frame: 8 years post-implant
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 88
Participants
  0 None | 58
  +1 Trivial | 20
  +2 Mild | 9
  +3 Moderate | 1
  +4 Severe | 0

15. Secondary Outcome: Subject's Average White Blood Cell Count Measurement Over Time.
Description: Laboratory analysis of White Blood Cell Count on blood drawn from subject; WBC fight infection.
Time Frame: 6 months and annually for 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliters
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
10^3 cells/microliters
  6 Months: number analyzed (Participants) | 221
  6 Months | 7.0 (2.0)
  1 Year: number analyzed (Participants) | 218
  1 Year | 6.8 (1.7)
  2 Years: number analyzed (Participants) | 203
  2 Years | 6.9 (1.7)
  3 Years: number analyzed (Participants) | 200
  3 Years | 6.9 (2.1)
  4 Years: number analyzed (Participants) | 189
  4 Years | 6.9 (2.1)
  5 Years: number analyzed (Participants) | 178
  5 Years | 6.9 (1.7)
  6 Years: number analyzed (Participants) | 169
  6 Years | 7.1 (2.3)
  7 Years: number analyzed (Participants) | 125
  7 Years | 7.2 (1.6)
  8 Years: number analyzed (Participants) | 88
  8 Years | 7.4 (2.3)

16. Secondary Outcome: Subject's Average Red Blood Cells Count Over Time.
Description: Laboratory Analysis of Red Blood Cell (RBC) Count on blood drawn from subjects; RBC carry oxygen.
Time Frame: 6 months and annually for 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliters
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
10^6 cells/microliters
  6 Months: number analyzed (Participants) | 220
  6 Months | 4.7 (0.6)
  1 Year: number analyzed (Participants) | 218
  1 Year | 4.7 (0.6)
  2 Years: number analyzed (Participants) | 203
  2 Years | 4.7 (0.5)
  3 Years: number analyzed (Participants) | 200
  3 Years | 4.6 (0.5)
  4 Years: number analyzed (Participants) | 189
  4 Years | 4.6 (0.5)
  5 Years: number analyzed (Participants) | 178
  5 Years | 4.6 (0.6)
  6 Years: number analyzed (Participants) | 169
  6 Years | 4.6 (0.5)
  7 Years: number analyzed (Participants) | 125
  7 Years | 4.7 (0.6)
  8 Years: number analyzed (Participants) | 88
  8 Years | 4.7 (0.5)

17. Secondary Outcome: Subject's Average Hematocrit Percentage Over Time.
Description: Laboratory Analysis of Hematocrit Percentage on blood drawn from subjects. Hematocrit is the proportion of red blood cells to the fluid component (plasma) in the blood.
Time Frame: 6 months and annually for 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
percentage of red blood cells
  6 Months: number analyzed (Participants) | 221
  6 Months | 40.6 (4.0)
  1 Year: number analyzed (Participants) | 218
  1 Year | 41.2 (4.0)
  2 Years: number analyzed (Participants) | 203
  2 Years | 41.7 (4.0)
  3 Years: number analyzed (Participants) | 200
  3 Years | 41.4 (3.9)
  4 Years: number analyzed (Participants) | 188
  4 Years | 41.8 (4.1)
  5 Years: number analyzed (Participants) | 177
  5 Years | 41.6 (7.9)
  6 Years: number analyzed (Participants) | 169
  6 Years | 41.2 (5.3)
  7 Years: number analyzed (Participants) | 125
  7 Years | 41.4 (4.6)
  8 Years: number analyzed (Participants) | 88
  8 Years | 42.6 (6.6)

18. Secondary Outcome: Subject's Average Hemoglobin Count Over Time.
Description: Laboratory Analysis of Hemoglobin Count on blood drawn from subjects. Hemoglobin is an oxygen-carrying protein in red blood cells.
Time Frame: 6 months and annually for 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
g/dl
  6 Months: number analyzed (Participants) | 221
  6 Months | 13.7 (1.6)
  1 Year: number analyzed (Participants) | 218
  1 Year | 14.0 (1.6)
  2 Years: number analyzed (Participants) | 203
  2 Years | 14.1 (1.6)
  3 Years: number analyzed (Participants) | 200
  3 Years | 14.0 (1.5)
  4 Years: number analyzed (Participants) | 189
  4 Years | 14.1 (1.5)
  5 Years: number analyzed (Participants) | 177
  5 Years | 14.0 (1.6)
  6 Years: number analyzed (Participants) | 169
  6 Years | 14.0 (1.7)
  7 Years: number analyzed (Participants) | 125
  7 Years | 14.0 (1.8)
  8 Years: number analyzed (Participants) | 88
  8 Years | 14.3 (1.4)

19. Secondary Outcome: Subject's Average Platelet Count Over Time.
Description: Laboratory Analysis of Platelet Count on blood drawn from subjects; platelets help with blood clotting.
Time Frame: 6 months and annually for 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 10^3 platelets per microliter
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
10^3 platelets per microliter
  6 Months: number analyzed (Participants) | 220
  6 Months | 207.9 (64.4)
  1 Year: number analyzed (Participants) | 218
  1 Year | 202.5 (50.1)
  2 Years: number analyzed (Participants) | 202
  2 Years | 204.7 (56.3)
  3 Years: number analyzed (Participants) | 200
  3 Years | 195.6 (50.9)
  4 Years: number analyzed (Participants) | 188
  4 Years | 198.6 (57.1)
  5 Years: number analyzed (Participants) | 178
  5 Years | 198.3 (74.7)
  6 Years: number analyzed (Participants) | 169
  6 Years | 196.9 (54.7)
  7 Years: number analyzed (Participants) | 125
  7 Years | 199.1 (58.3)
  8 Years: number analyzed (Participants) | 88
  8 Years | 190.7 (51.1)

20. Secondary Outcome: Subject's Average Serum Lactate Dehydrogenase (LDH) Over Time.
Description: Laboratory Analysis of Serum Lactate Dehydrogenase on blood drawn from subjects; The lactate dehydrogenase (LDH) test looks for signs of damage to the body's tissues.
Time Frame: 6 months and annually for 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
U/L
  6 Months: number analyzed (Participants) | 216
  6 Months | 240.8 (112.6)
  1 Year: number analyzed (Participants) | 217
  1 Year | 235.5 (103.3)
  2 Years: number analyzed (Participants) | 198
  2 Years | 234.6 (106.5)
  3 Years: number analyzed (Participants) | 197
  3 Years | 236.1 (102.3)
  4 Years: number analyzed (Participants) | 187
  4 Years | 243.9 (107.1)
  5 Years: number analyzed (Participants) | 171
  5 Years | 236.7 (94.3)
  6 Years: number analyzed (Participants) | 168
  6 Years | 255.3 (162.2)
  7 Years: number analyzed (Participants) | 122
  7 Years | 238.2 (88.5)
  8 Years: number analyzed (Participants) | 86
  8 Years | 263.0 (117.9)

21. Secondary Outcome: Subject's Average Haptoglobin Measurement Over Time.
Description: Laboratory Analysis of haptoglobin on blood drawn from subjects; haptoglobin is a protein produced by the liver.
Time Frame: 6 months and annually for 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
mg/dl
  6 Months: number analyzed (Participants) | 204
  6 Months | 118.4 (66.9)
  1 Year: number analyzed (Participants) | 203
  1 Year | 114.7 (70.7)
  2 Years: number analyzed (Participants) | 188
  2 Years | 115.6 (61.4)
  3 Years: number analyzed (Participants) | 181
  3 Years | 116.3 (58.9)
  4 Years: number analyzed (Participants) | 169
  4 Years | 112.8 (62.3)
  5 Years: number analyzed (Participants) | 159
  5 Years | 127.1 (104.0)
  6 Years: number analyzed (Participants) | 154
  6 Years | 115.6 (58.9)
  7 Years: number analyzed (Participants) | 107
  7 Years | 125.0 (87.4)
  8 Years: number analyzed (Participants) | 80
  8 Years | 109.8 (53.7)

22. Secondary Outcome: Subject's Average Reticulocytes Percentage Over Time.
Description: Laboratory Analysis of reticulocytes on blood drawn from subjects. Reticulocytes are newly produced immature red blood cells; a reticulocyte blood test measures the amount of these cells in the blood.
Time Frame: 6 months and annually for 8 years post-implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of reticulocytes
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 258
percentage of reticulocytes
  6 Months: number analyzed (Participants) | 214
  6 Months | 1.2 (1.5)
  1 Year: number analyzed (Participants) | 214
  1 Year | 1.2 (0.5)
  2 Years: number analyzed (Participants) | 199
  2 Years | 1.2 (0.5)
  3 Years: number analyzed (Participants) | 196
  3 Years | 1.2 (0.5)
  4 Years: number analyzed (Participants) | 186
  4 Years | 1.4 (1.3)
  5 Years: number analyzed (Participants) | 170
  5 Years | 1.8 (6.2)
  6 Years: number analyzed (Participants) | 168
  6 Years | 4.4 (13.4)
  7 Years: number analyzed (Participants) | 121
  7 Years | 5.4 (16.5)
  8 Years: number analyzed (Participants) | 84
  8 Years | 4.5 (14.8)

23. Secondary Outcome: Subject's Average Score on the EQ-5D- Quality of Life Questionnaire at Baseline and 6 Months Post-Implant.
Description: The EQ-5D is a standardized questionnaire that asks subjects to rate themselves (no problems, some problems, extreme problems) on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale ranges from a minimum of 0 and a maximum of 100 where zero is the 'worst state imaginable' and 100 is the 'best state imaginable'.
Time Frame: Baseline and 6 Months Post-Implant
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
Number analyzed (Participants) | 96
units on a scale
  Baseline | 75.8 (15.1)
  6 Months Follow-up | 84.3 (13.6)

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through eight years post implant.
Description: The outcome is reported for subjects who received the Carpentier-Edwards PERIMOUNT Magna Ease Pericardial Bioprosthesis, Model 3300TFX device where data is available.
Arm/Group | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX
All-Cause Mortality (participants affected / at risk) | 38/258
Serious Adverse Events (participants affected / at risk) | 211/258
Other Adverse Events (participants affected / at risk) | 184/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX (N=258)
Anemia (Blood and lymphatic system disorders) | 20 (23)
Angina (Cardiac disorders) | 11 (16)
Arrhythmia (Cardiac disorders) | 87 (101)
Bleeding - Major (Blood and lymphatic system disorders) | 32 (34)
Bleeding - Minor (Blood and lymphatic system disorders) | 12 (12)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 9 (9)
Cancer (General disorders) | 27 (39)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Cardiac Conduction Disturbance (Cardiac disorders) | 6 (6)
Cardiac Failure (Cardiac disorders) | 14 (17)
Cardiovascular - Other (Cardiac disorders) | 11 (11)
Cardiovascular Dissection / Tear / Injury (Cardiac disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Drug Reaction (General disorders) | 3 (3)
Edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Endocarditis (Cardiac disorders) | 6 (6)
Fever - Unknown Origin (General disorders) | 2 (3)
Gastro-Intestinal Complication (Gastrointestinal disorders) | 26 (32)
Hematological Disorder (Blood and lymphatic system disorders) | 6 (8)
Hepatic Complication (Gastrointestinal disorders) | 3 (3)
Hypotension (Cardiac disorders) | 2 (2)
Infection / Inflammation (Infections and infestations) | 40 (54)
Metabolic Complication (Metabolism and nutrition disorders) | 3 (3)
Mitral Regurgitation (Native) (Cardiac disorders) | 1 (1)
Multiple Organ Failure (General disorders) | 5 (5)
Myocardial Infarct (Cardiac disorders) | 7 (7)
NSVD - Other non-structural valve dysfunction (Cardiac disorders) | 1 (1)
NSVD - Paravalvular Leak - Major (Cardiac disorders) | 2 (2)
NSVD - Paravalvular Leak - Minor (Cardiac disorders) | 1 (1)
Neurological Complication (Psychiatric disorders) | 8 (8)
Other (General disorders) | 63 (99)
Pericardial Effusion (Cardiac disorders) | 20 (21)
Pleural Effusion (Cardiac disorders) | 37 (37)
Pneumothorax / Hemothorax (Cardiac disorders) | 1 (1)
Psychiatric Complication (Psychiatric disorders) | 6 (6)
Pulmonary Embolism (Cardiac disorders) | 3 (3)
Renal Complication (Renal and urinary disorders) | 6 (6)
Respiratory Complication (Respiratory, thoracic and mediastinal disorders) | 27 (30)
SVD - Other structural valve deterioration (Cardiac disorders) | 8 (8)
SVD - Study valve calcification (Cardiac disorders) | 2 (2)
Septicemia (Blood and lymphatic system disorders) | 5 (7)
Sternal / Thoracic Wound Complication (Musculoskeletal and connective tissue disorders) | 9 (12)
Sudden Death (General disorders) | 2 (2)
Syncope (Cardiac disorders) | 2 (3)
Thromboembolism - Non-cerebral (Cardiac disorders) | 1 (1)
Thromboembolism - Stroke (Cardiac disorders) | 13 (13)
Thromboembolism - TIA (Cardiac disorders) | 6 (6)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3)
Vascular Complication (Cardiac disorders) | 9 (13)
Vision Disorder (Eye disorders) | 8 (10)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carpentier-Edwards® PERIMOUNT® Magna Ease™, Model 3300TFX (N=258)
Abnormal Lab Values (Eye disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Angina (Cardiac disorders) | 4 (6)
Arrhythmia (Cardiac disorders) | 58 (80)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bleeding - Minor (Blood and lymphatic system disorders) | 12 (13)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 7 (7)
Cancer (General disorders) | 4 (4)
Cardiac Conduction Disturbance (Cardiac disorders) | 15 (15)
Cardiac Failure (Cardiac disorders) | 2 (2)
Cardiovascular - Other (Cardiac disorders) | 7 (8)
Drug Reaction (General disorders) | 1 (1)
Edema (Musculoskeletal and connective tissue disorders) | 2 (2)
Fever - Unknown Origin (General disorders) | 5 (5)
Gastro-Intestinal Complication (Gastrointestinal disorders) | 10 (10)
Hematological Disorder (Blood and lymphatic system disorders) | 3 (4)
Hemolysis (Cardiac disorders) | 2 (2)
Hepatic Complication (Hepatobiliary disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Infection / Inflammation (Infections and infestations) | 42 (48)
Metabolic Complication (Metabolism and nutrition disorders) | 1 (1)
Myocardial Infarct (Cardiac disorders) | 2 (2)
NSVD - Paravalvular Leak - Minor (Cardiac disorders) | 1 (1)
Neurological Complication (Nervous system disorders) | 1 (1)
Other (General disorders) | 84 (165)
Pericardial Effusion (Cardiac disorders) | 17 (17)
Pleural Effusion (Cardiac disorders) | 36 (37)
Pneumothorax / Hemothorax (Cardiac disorders) | 3 (3)
Psychiatric Complication (Psychiatric disorders) | 2 (2)
Pulmonary Embolism (Cardiac disorders) | 1 (1)
Renal Complication (Renal and urinary disorders) | 6 (7)
Respiratory Complication (Respiratory, thoracic and mediastinal disorders) | 15 (17)
SVD - Other structural valve deterioration (Cardiac disorders) | 5 (5)
Septicemia (Blood and lymphatic system disorders) | 1 (1)
Sternal / Thoracic Wound Complication (Musculoskeletal and connective tissue disorders) | 3 (3)
Syncope (Cardiac disorders) | 7 (7)
Thromboembolism - Non-cerebral (Cardiac disorders) | 1 (1)
Thromboembolism - TIA (Cardiac disorders) | 5 (5)
Tricuspid Regurgitation (Native) (Cardiac disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 2 (3)
Vascular Complication (Cardiac disorders) | 4 (4)
Vision Disorder (Eye disorders) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of overall study results which have not been released requires written approval of Sponsor, but presentation of site-specific results can occur subject to review by Sponsor. Manuscripts will be submitted to Sponsor for review 60 days prior to submission of manuscript for publication/presentation. Sponsor may ask for a 90 day delay of submission of manuscripts for publication to protect proprietary information and filing of related patent applications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-09-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT01171625/Prot_SAP_000.pdf